CLINICAL TRIAL: NCT05306496
Title: Laparoscopic Inguinal and Femoral heRniA rePaIr Using Pre-shapeD 4DMESH® (4DLap): Assessing Hernia Recurrence and Pain up to 5-years Follow-up
Brief Title: Laparoscopic Inguinal and Femoral heRniA rePaIr Using Pre-shapeD 4DMESH® (4DLap)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cousin Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPID4D
Record Dates: First submitted 2022-02-24; First posted 2022-04-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Inguinal Hernia; Femoral Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pre-shaped 4DMESH® — The 4DMESH® mesh is semi-resorbable parietal reinforcement implant made of 25% Polypropylene (non-resorbable) and 75% Poly-L-Lactic Acid (resorbable). 4DMESH® meshes are designed for the repair and reinforcement of inguinal and femoral hernias. 4DMesh is a CE-marked, class III medical device manufactured by Cousin Biotech.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the 4DMESH® used in (robot-assisted) laparoscopic inguinal and femoral hernia repair. The goal of the study will be achieved by assessing the prevalence of recurrences, pain, quality-of-life (QoL), return to daily activities and work and groin symptoms, and by reporting of peri- and postoperative complications in a prospectively maintained database.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a primary unilateral or primary bilateral inguinal or femoral hernia eligible for (robot-assisted) laparoscopic TEP or TAPP repair.
2. Patients with American Society of Anesthesiologists (ASA) grade I to III.
3. Patient ≥ 18 years of age at study entry.
4. Patient and investigator signed and dated the informed consent form prior to the index-procedure.

Exclusion Criteria:

1. Patient has a recurrent inguinal or femoral hernia.
2. Patient is treated using the Lichtenstein technique.
3. Patients with ASA grade IV and V.
4. Patient is allergic to the components of the 4DMESH®.
5. Presence of an infected site.
6. Patient has a life expectancy of less than 5 years.
7. Patient is unable / unwilling to provide informed consent.
8. Patient is unable to comply with the protocol or proposed follow-up visits.
9. Patient is enrolled in another study (BE/ES) / Participation in a clinical trial within 3 months prior to the initial visit (FR).
10. Patient is pregnant (BE/FR) / Pregnant women (ES).
11. Patient benefiting from a legal protection measure (minors, under guardianship, curatorship, safeguard of justice, future protection mandate or family empowerment) (FR).
12. Patient not benefiting from a social protection scheme (FR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | At 12-months follow-up
  To determine the prevalence of hernia recurrence at 12-months follow-up via an abdominal ultrasound during an in-hospital visit.

SECONDARY OUTCOMES:
Technical success | At index-procedure
  To determine the percentage of procedures with technical success, defined as (robot-assisted) laparoscopic TEP or TAPP as intended without technical difficulties and without conversion to open laparotomy.
Duration of surgery | At index-procedure
  To determine the mean duration of the surgery.
Duration of hospital stay | At the moment the patient is discharged from the hospital after the procedure (discharge), an average of 1 day
  To determine the mean duration of hospital stay.
Peri- and post-operative complications related to 4DMESH® | At 5-years follow-up
  To determine the rate of peri- and post-operative complications related to 4DMESH® up to 5-years follow-up.
Early recurrences | At 4-5 weeks follow-up
  To determine the early recurrence rate at 4-5 weeks follow-up.
Late recurrence rate | At 24-months follow-up
  To determine the recurrence rate at 24-months follow-up (Patient Reported Outcome Measure (PROM) via telephone call).
Late recurrence rate | At 60-months follow-up
  To determine the recurrence rate at 60-months follow-up (Patient Reported Outcome Measure (PROM) via telephone call).
Mesh migration and mesh shrinkage | At 12-months follow-up
  To evaluate the incidence of mesh migration and mesh shrinkage at 12-months follow-up via abdominal ultrasound (only in specialized investigational centers ).
Re-intervention | At 5-years follow-up
  To determine the incidence of hernia surgery related re-interventions since the (robot-assisted) laparoscopic TEP or TAPP procedure.
Explantation rate | At 5-years follow-up
  To determine the explantation rate since the (robot-assisted) laparoscopic TEP or TAPP procedure.
Return to daily activities | At 4-5 weeks follow-up
  To determine the mean number of days when the patient returned to daily activities after the operation, assessed at 4-5 weeks follow-up.
Return to work | At 4-5 weeks follow-up
  To determine the mean number of days when the patient returned to work after the operation, assessed at 4-5 weeks follow-up.
Pre-operative pain scoring | At baseline
  To determine pain (at rest, normal activity, strenuous activity) assessed using the McCarthy visual analogue scale (0-150 mm, higher score means more pain).
Post-operative pain scoring | At discharge, an average of 1 day
  To determine pain (at rest, normal activity, strenuous activity) assessed using the McCarthy visual analogue scale (0-150 mm, higher score means more pain).
Post-operative pain scoring | At 4-5 weeks follow-up
  To determine pain (at rest, normal activity, strenuous activity) assessed using the McCarthy visual analogue scale (0-150 mm, higher score means more pain).
Post-operative pain scoring | At 12-months follow-up
  To determine pain (at rest, normal activity, strenuous activity) assessed using the McCarthy visual analogue scale (0-150 mm, higher score means more pain).
Post-operative pain scoring | At 24-months follow-up
  To determine pain (at rest, normal activity, strenuous activity) assessed using the McCarthy visual analogue scale (0-150 mm, higher score means more pain).
Post-operative pain scoring | At 60-months follow-up
  To determine pain (at rest, normal activity, strenuous activity) assessed using the McCarthy visual analogue scale (0-150 mm, higher score means more pain).
Intake of analgesics | At the moment the patient is discharged from the hospital after the procedure (discharge), an average of 1 day
  To register intake of analgesics.
Intake of analgesics | At 4-5 weeks follow-up
  To register intake of analgesics.
Intake of analgesics | At 12-months follow-up
  To register intake of analgesics.
Intake of analgesics | At 24-months follow-up
  To register intake of analgesics.
Intake of analgesics | At 60-months follow-up
  To register intake of analgesics.
QoL | At baseline
  To assess QoL by the EQ-5D questionnaire.
QoL | At 4-5 weeks follow-up
  To assess QoL by the EQ-5D questionnaire.
QoL | At 12-months follow-up
  To assess QoL by the EQ-5D questionnaire.
QoL | At 24-months follow-up
  To assess QoL by the EQ-5D questionnaire.
QoL | At 60-months follow-up
  To assess QoL by the EQ-5D questionnaire.
EQ-5D change | At 4-5 weeks follow-up
  To determine EQ-5D change assessed by minimally important differences at baseline and follow-up (outcome: worse, no change, better).
EQ-5D change | At 12-months follow-up
  To determine EQ-5D change assessed by minimally important differences at baseline and follow-up (outcome: worse, no change, better).
EQ-5D change | At 24-months follow-up
  To determine EQ-5D change assessed by minimally important differences at baseline and follow-up (outcome: worse, no change, better).
EQ-5D change | At 60-months follow-up
  To determine EQ-5D change assessed by minimally important differences at baseline and follow-up (outcome: worse, no change, better).
Subjective groin symptoms | At 4-5 weeks follow-up
  To assess the occurrence of subjective groin symptoms at follow-up (awareness of groin lump, perception of foreign material in groin, loss of skin sensation in groin, discomfort in groin).
Subjective groin symptoms | At 12-months follow-up
  To assess the occurrence of subjective groin symptoms at follow-up (awareness of groin lump, perception of foreign material in groin, loss of skin sensation in groin, discomfort in groin).
Subjective groin symptoms | At 24-months follow-up
  To assess the occurrence of subjective groin symptoms at follow-up (awareness of groin lump, perception of foreign material in groin, loss of skin sensation in groin, discomfort in groin).
Subjective groin symptoms | At 60-months follow-up
  To assess subjective groin symptoms at follow-up (awareness of groin lump, perception of foreign material in groin, loss of skin sensation in groin, discomfort in groin).
Global groin symptoms | At 4-5 weeks follow-up
  To assess the level of global groin symptoms at follow-up compared to baseline (outcome: worse, no change, better).
Global groin symptoms | At 12-months follow-up
  To assess the level of global groin symptoms at follow-up compared to baseline (outcome: worse, no change, better).
Global groin symptoms | At 24-months follow-up
  To assess the level of global groin symptoms at follow-up compared to baseline (outcome: worse, no change, better).
Global groin symptoms | At 60-months follow-up
  To assess the level of global groin symptoms at follow-up compared to baseline (outcome: worse, no change, better).
Impact on sex life | At 4-5 weeks follow-up
  To assess the impact on sex life at follow-up compared to baseline (outcome: worse, no change, better).
Impact on sex life | At 12-months follow-up
  To assess the impact on sex life at follow-up compared to baseline (outcome: worse, no change, better).
Impact on sex life | At 24-months follow-up
  To assess the impact on sex life at follow-up compared to baseline (outcome: worse, no change, better).
Impact on sex life | At 60-months follow-up
  To assess the impact on sex life at follow-up compared to baseline (outcome: worse, no change, better).

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (3):
  - Ziekenhuis Oost-Limburg Genk, Genk, Limburg
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen, Vlaams-Brabant
  - AZ Groeninge, Kortrijk, West-Vlaanderen
- France (4):
  - Hôpital Lyon Sud, Hospices Civils de Lyon, Lyon
  - CHU de Nantes, Nantes
  - CHU de Reims, Reims
  - CH de Tourcoing, Tourcoing
- Spain (2):
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Viamed Santa Ángela de la Cruz en Sevilla, Seville

IPD SHARING:
Plan to Share IPD: No